CLINICAL TRIAL: NCT02241720
Title: Regorafenib as a Second Line Single Agent in the Treatment of Metastatic or Advanced Adenocarcinoma of the Esophagus, Gastroesophageal Junction or Stomach
Brief Title: Regorafenib Second Line Treatment of Metastatic or Advanced Upper GI Cancers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI68135
Record Dates: First submitted 2013-11-21; First posted 2014-09-16 (Estimated); Results first posted 2017-10-26 (Actual); Last update posted 2018-01-11 (Actual); Status verified 2017-12

CONDITIONS: Upper GI Cancer
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Regorafenib treatment (Experimental)
  Interventions: Drug: regorafenib

INTERVENTIONS:
Drug: regorafenib

SUMMARY:
Regorafenib as a Second Line Single Agent in the Treatment of Metastatic or Advanced Adenocarcinoma of the Esophagus, Gastroesophageal Junction or Stomach

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of metastatic or locally advanced inoperable adenocarcinoma of the esophagus, gastroesophageal junction or stomach.
* Patients must show signs of progression during or less than 4 months after being treated with a first line therapy for their metastatic or locally advanced inoperable cancer.
* Patients must have measureable disease at screening by Response Evaluation Criteria for Solid Tumors 1.1 criteria
* Age greater than or equal to 18 years.
* Eastern Cooperative Oncology Group Performance Status 0-1
* Subjects must be able to understand and be willing to sign the written informed consent form. A signed informed consent form must be appropriately obtained prior to the conduct of any trial-specific procedure.
* All acute toxic effects of any prior treatment have resolved to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 Grade 1 or less at the time of signing the Informed Consent Form. Alopecia (any grade) and peripheral neuropathy less than grade 2 is allowed.
* Adequate bone marrow, liver and liver function as assessed by laboratory requirement
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of study drug. Post-menopausal women (defined as no menses for at least 1 year) and surgically sterilized women are not required to undergo a pregnancy test.
* Subjects (men and women) of childbearing potential must agree to use adequate contraception beginning at the signing of the informed consent form until at least 3 months after the last dose of study drug. Highly effective contraception must be used (male condom with spermicidal, diaphragm with spermicidal, intra-uterine device) by both sexes.
* Subject must be able to swallow and retain oral medication.

Exclusion Criteria:

* Prior use of regorafenib
* Uncontrolled hypertension (systolic pressure greater than 140 mm Hg or diastolic pressure greater than 90 mm Hg National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 on repeated measurement) despite optimal medical management.
* Active or clinically significant cardiac disease including:
* Congestive heart failure - New York Heart Association greater than Class 2.
* Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers.
* Unstable angina (anginal symptoms at rest), new-onset angina within 3 months before randomization, or myocardial infarction within 6 months before randomization.
* Evidence or history of bleeding diathesis or coagulopathy.
* Any hemorrhage or bleeding event greater than or equal to National Cancer Institute Common Terminology Criteria for Adverse Events Grade 3 within 4 weeks prior to start of study medication.
* Subjects with thrombotic, embolic, venous, or arterial events, such as cerebrovascular accident (including transient ischemic attacks) deep vein thrombosis or pulmonary embolism within 6 months of start of study treatment
* Subjects with any previously untreated or concurrent cancer that is distinct in primary site or histology except cervical cancer in-situ, treated basal cell carcinoma, or superficial bladder tumor. Subjects surviving a cancer that was curatively treated and without evidence of disease for more than 3 years before randomization are allowed. All cancer treatments must be completed at least 3 years prior to start of study treatment.
* Patients with severe hepatic impairment (Child-Pugh Class C)
* Known history of human immunodeficiency virus infection or current chronic or active hepatitis B or C infection requiring treatment with antiviral therapy.
* Patients requiring intravenous antiviral or intravenous antibiotic treatment for ongoing infections
* Symptomatic metastatic brain or meningeal tumors.
* Presence of a non-healing wound, non-healing skin ulcer, or bone fracture.
* Patient's with a history of kidney disease or persistent proteinuria must have less than Grade 3 proteinuria per NCI CTCAE v4.0 at screening. If a patient has a history of kidney disease or persistent proteinuria, a urine protein test will be performed on a random urine sample. If the result is normal then no additional testing is required. If the result is abnormal, a 24 hour urine will be collected to determine if proteinuria is less than Grade 3.
* Interstitial lung disease with ongoing signs and symptoms at the time of informed consent.
* Pleural effusion or ascites that causes respiratory compromise (greater than or equal to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 Grade 2 dyspnea). Patients may undergo thoracentesis and paracentesis to improve symptoms prior to enrollment.
* History of organ allograft (including corneal transplant).
* Known or suspected grade 3 allergy or hypersensitivity to any of the study drugs, study drug classes, or excipients of the formulations given during the course of this trial.
* Any malabsorption condition that in the opinion of the investigator would significantly impact drug absorption.
* Women who are pregnant or breast-feeding.
* Any condition which, in the investigator's opinion, makes the subject unsuitable for trial participation.
* Substance abuse, medical, psychological or social conditions that in the opinion of the investigator may interfere with the subject's participation in the study or evaluation of the study results.
* Concurrent anti-cancer therapy (chemotherapy, radiation therapy, surgery, immunotherapy, biologic therapy, or tumor embolization) within 28 days of starting study treatment. Palliative radiation is allowed.
* Concurrent use of another investigational drug or device during, or within 3 weeks of starting study treatment.
* Concurrent use of strong CYP3A4 inducers (e.g. rifampin, phenytoin, carbamazepine, phenobarbital, and St. John's Wort)
* Concurrent use with strong inhibitors of CYP3A4 (e.g. clarithromycin, grapefruit juice, itraconazole, ketoconazole, nefazadone, posaconazole, telithromycin, and voriconazole)
* Major surgical procedure, open biopsy, or significant traumatic injury within 3 weeks before start of study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Regorafenib Treatment: 160 mg regorafenib by mouth once daily for 3 weeks of every 4 week cycle
Period: Overall Study
Arm/Group | Regorafenib Treatment
Started | 5
Completed | 1
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- Regorafenib Treatment: regorafenib
Arm/Group | Regorafenib Treatment
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Stable Disease at Eight Weeks Post-Treatment
Description: Patients had disease assessed by CT scans. Stable Disease is defined by any response better than Progression as defined by RECIST 1.1. Progression is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 5 months - 3 months treatment and 8 weeks post end of treatment visit
Population: 3 subjects did not complete an 8 week EOT visit for: Death, Patient W/D, AE.
Measure: Count of Participants; unit: Participants
Arm/Group | Regorafenib Treatment
Number analyzed (Participants) | 2
Participants | 2

ADVERSE EVENTS:
Arm/Group | Regorafenib Treatment
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib Treatment (N=5)
Disease Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
heart failure (Cardiac disorders) | 1 (1)
Tracheoesophageal fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib Treatment (N=5)
Fatigue (General disorders) | 3 (3)
Hypertension (Vascular disorders) | 4 (4)
deydration (Metabolism and nutrition disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
hyperbilirubinemia (Investigations) | 1 (1)
maculopapular rash (Skin and subcutaneous tissue disorders) | 1 (2)
anemia (Blood and lymphatic system disorders) | 1 (1)
hypothyroidism (Endocrine disorders) | 1 (1)
dysphagia (Gastrointestinal disorders) | 2 (2)
headache (Nervous system disorders) | 1 (1)
oral pain (Gastrointestinal disorders) | 1 (1)
mucositis oral (Gastrointestinal disorders) | 2 (2)
syncope (Nervous system disorders) | 1 (1)
hypotension (Vascular disorders) | 1 (1)
voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No